CLINICAL TRIAL: NCT06237387
Title: Association of Acne Vulgaris With Oral Hygiene and Severity of Plaque-Induced Gingivitis in Puberty
Brief Title: Association of Acne Vulgaris With Oral Hygiene and Gingivitis
Status: Not yet recruiting | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Okumuş, Assistant Professor, Erzincan University
Other Study IDs: EUDF-OKUMUS-003
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Acne Vulgaris; Gingivitis; Dental Plaque; Oral Hygiene; Puberty
MeSH Terms: conditions — Acne Vulgaris; Gingivitis; Dental Plaque

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients with Allen-Smith acne score 0 and 2 (Mild lesions)
  Interventions: Other: Periodontal examination
- Group B: Patients with Allen-Smith acne score 4 (Moderate lesions)
  Interventions: Other: Periodontal examination
- Group C: Patients with Allen-Smith acne score 6 and 8 (Severe lesions)
  Interventions: Other: Periodontal examination

INTERVENTIONS:
Other: Periodontal examination — Determining the patient's oral hygiene status and the severity of gingivitis. For this purpose, the non-invasive Löe-Silness plaque and gingival index system will be used.

SUMMARY:
The goal of this observational study is to learn about in the relationship between acne vulgaris and oral hygiene and gingivitis. The main questions it aims to answer are:

* Is there a relationship between the severity of acne vulgaris lesions and the severity of plaque-related gingivitis?
* Could oral hygiene or the severity of plaque-related gingivitis have an impact on the treatment of acne lesions?

Participants will;

* First be examined at the dermatology clinic.
* Then be examined at the periodontology clinic.
* Participants with severe acne vulgaris lesions will be examined a second time at the dermatology clinic. (1.5 months after the first examination)
* Regularly use the antibiotic containing 100 mg doxycycline prescribed in the dermatology clinic for acne treatment. (Patients deemed suitable by the dermatologist)

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy
* Not using any medication regularly
* Not having received acne treatment before
* Not having a known allergy to Doxycycline/Tetracycline antibiotics
* Not having received periodontal disease treatment in the last 6 months
* Not having taken antibiotics or anti-inflammatory drugs in the last month
* Not having used antiseptic mouthwash in the last month
* Being between the ages of 13-18
* No radiographic bone loss or clinical attachment loss
* Absence of any diagnosed psychiatric disease

Exclusion Criteria:

* Smoking
* Using antibiotics and anti-inflammatory drugs
* Having significant psychological problems
* Mouth breathing

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants in puberty between the ages of 13-18.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-05 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
The relationship between acne vulgaris and the severity of gingivitis depending on the amount of plaque | Baseline
  Data from three groups will be presented as the correlation between the Gingival Index score and the Plaque Index score. The relationship between the severity of gingival inflammation depending on the amount of plaque and acne lesions will be evaluated.
The relationship between acne vulgaris and oral hygiene | Baseline
  Describes the relationship between plaque index data obtained during periodontal examination of patients and acne lesions.
  According to the plaque index system, a score of "0" indicates the absence of plaque. A score of "1" refers to the amount of plaque that is not visible to the eye but detected by the periodontal probe. A score of "2" refers to the amount of plaque detectable visually. The highest score, "3", indicates excessive plaque accumulation.
Relationship between acne vulgaris and gingival index | Baseline
  To compare gingival index values obtained during periodontal examination with acne vulgaris, regardless of plaque index values.
  According to the gingival index system, a score of "0" indicates completely healthy gums. A score of "1" indicates mild erythema and no bleeding on probing. A score of "2" indicates a small amount of bleeding on probing. The highest score, "3", indicates spontaneous or excessive gingival bleeding.

SECONDARY OUTCOMES:
The relationship between response to medical treatment and severity of gingivitis depending on the amount of plaque | At the end of 1.5 months from the beginning
  The relationship between the response to medical treatment at the end of 1.5 months from the beginning and the severity of gingivitis depending on the amount of plaque in Group C (severe periodontitis) patients
The relationship between response to medical treatment and oral hygiene | At the end of 1.5 months from the beginning
  Response to medical treatment in Group C (severe periodontitis) patients at the end of 1.5 months from the beginning. The relationship between response to medical treatment and plaque index.
  According to the plaque index system, a score of "0" indicates the absence of plaque. A score of "1" refers to the amount of plaque that is not visible to the eye but detected by the periodontal probe. A score of "2" refers to the amount of plaque detectable visually. The highest score, "3", indicates excessive plaque accumulation.
The relationship between response to medical treatment and gingival index | At the end of 1.5 months from the beginning
  Response to medical treatment in Group C (severe periodontitis) patients after 1.5 months from the beginning. The relationship between response to medical treatment and gingival index.
  According to the gingival index system, a score of "0" indicates completely healthy gums. A score of "1" indicates mild erythema and no bleeding on probing. A score of "2" indicates a small amount of bleeding on probing. The highest score, "3", indicates spontaneous or excessive gingival bleeding.